CLINICAL TRIAL: NCT05248919
Title: Therapy for Hepatitis C Virus (HCV) in Primary Treatment Failure in Pakistan
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Aga Khan University (Other); Dow University of Health Sciences (Other); University of Oxford (Other); University of Bristol (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCVTreatmentFailure
Record Dates: First submitted 2021-06-30; First posted 2022-02-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination; Sofosbuvir; velpatasvir

STUDY DESIGN:
Intervention Model Description: 268 patients accepted into the study will be divided into two groups (134 per group) and randomly allocated 1:1 (stratified by the presence or absence of cirrhosis) to receive: i) 12 weeks treatment with sofosbuvir/velpatasvir or ii) 24 weeks treatment with sofosbuvir/velpatasvir. Approximately an additional 50 patients with decompensated cirrhosis will form the observational group iii) who will receive 24 weeks of sofosbuvir/velpatasvir. Patients will be assessed for sustained virological response (SVR) from the point of randomisation at 12 (+/-1 week) and 24 weeks (+/-1 week) and then finally at 36 weeks (+/-2 weeks).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 12 weeks - treatment with sofosbuvir/velpatasvir (usual regime) (Active Comparator): 134 first-line treatment failure patients randomly allocated to receive 12 weeks treatment with sofosbuvir/velpatasvir. 1:1 random allocation with stratification for the presence of cirrhosis
  Interventions: Drug: Epclusa (nucleotide HCV NS5B polymerase inhibitors).
- 24 weeks - treatment with sofosbuvir/velpatasvir (intervention) (Active Comparator): 134 first-line treatment failure patients randomly allocated to receive 24 weeks treatment with sofosbuvir/velpatasvir. 1:1 random allocation with stratification for the presence of cirrhosis
  Interventions: Drug: Epclusa (nucleotide HCV NS5B polymerase inhibitors).
- Observational (No Intervention): 50 patients with decompensated cirrhosis who will receive 24 weeks of sofosbuvir/velpatasvir.

INTERVENTIONS:
Drug: Epclusa (nucleotide HCV NS5B polymerase inhibitors). — Sofosbuvir (400mg/day) and Velpatasvir(100mg/day) for 12 weeks or 24 weeks
  Other Names: Sofosbuvir 400 Mg and Velpatasvir 100 Mg Oral Capsules
  Arms: 12 weeks - treatment with sofosbuvir/velpatasvir (usual regime); 24 weeks - treatment with sofosbuvir/velpatasvir (intervention)

SUMMARY:
This trial is linked to a largescale observational study determining the efficacy of sofosbuvir/daclatasvir in people in Pakistan (involving a separate protocol). The observational study will identify a cohort of patients who have not responded to first-line antiviral therapy (sofosbuvir plus daclatasvir) and the optimal treatment for these patients is unclear. This trial will address this issue by comparing two second-line treatment regimens to determine the preferred treatment option.

DETAILED DESCRIPTION:
Chronic infection with the hepatitis C virus (HCV) causes liver damage and, in many, liver cancer. We have effective drugs allowing us to cure most infected people and this stops the liver becoming damaged. Hepatitis C is common in Pakistan and the government is planning a massive national program to find and treat everyone who is infected. The government funded treatment program will fund therapy and assumes that the drugs will cure the vast majority of infected people and hence, in line with international recommendations, they are not planning to evaluate treatment outcomes. The efficacy of the drugs used in Pakistan (sofosbuvir plus daclatasvir) have not been widely assessed in the Pakistani population and their efficacy is not yet proven. In a separate protocol the efficacy of first line therapy in Pakistan will be determined and this study will examine the optimal management for people who have not responded.

This trial will determine optimal treatment regimens in resource poor settings by comparing two affordable, readily available treatment options. 268 patients who meet the inclusion criteria and who accept participation will be enrolled. These patients will be randomly allocated to two equal sized groups (134 per group) and allocated 1:1 (stratified by the presence or absence of cirrhosis) to receive: i) 12 weeks treatment with sofosbuvir/velpatasvir or ii) 24 weeks treatment with sofosbuvir/velpatasvir. An additional 50 patients with decompensated cirrhosis will form a third observational group iii) who will receive 24 weeks of sofosbuvir/velpatasvir. Patients will be assessed for sustained virological response (SVR) from the point of randomisation at 12 (+/-1 week) and 24 weeks (+/-1 week) and then finally at 36 weeks (+/-2 weeks).

The study outline is as follows:

1) HCV patients who fail to respond to the first-line therapy regime will be identified via sustained virological response (SVR) assessment 12 weeks (range 11-18 weeks) after completion of a course of all oral antiviral therapy with sofosbuvir plus daclatasvir for either 12 or 24 weeks with or without ribavirin provided by a recognized provider of health care in Pakistan.

* Potential participants who have been invited to participate will have a member of the medical team explain the details of the trial, they will then be given a maximum of 24h to read the relevant information sheets and to speak to a clinical member of the study team to ask any further questions, before they commence the process of fully informed consent.
* After obtaining written informed consent, a study specific participant identification number (ID) will be assigned to the participant.
* Consenting patients will have venepuncture performed as per the site's standard operating procedure (SOP). The donated pre-treatment plasma sample will be retained
* Once enrolled, the 268 patients accepted into the study will be randomly allocated into two groups (134 patients per group) using a computerised 1:1 randomisation programme (stratified by the presence or absence of decompensated cirrhosis) to receive:

  i) sofosbuvir(400mg/day)/velpatasvir (100mg/day) - 12 weeks ii) sofosbuvir(400mg/day)/velpatasvir (100mg/day) - 24 weeks
* The third observational group of decompensated patients (up to 50 patients) will be given sofosbuvir (400mg/day)/velpatasvir (100mg/day) - 24 weeks
* All patients will be treated for either 12 or 24 weeks.
* Each patient will be reviewed at weeks: 4 (+/- 1 week), 12 (+/-1 week), 24 (+/-1 week) and 36 ((+/- 2 week) after the first dose of second-line treatment (randomisation).
* Patients with second-line treatment failure will have 10ml blood sample taken for viral sequencing.
* Data will be collected on paper case report forms (CRFs) which will be securely stored prior to the data being transferred to a secure on-line database. Paper records will be retained as primary source documents.
* Cost effectiveness of the treatment regimens will be measured from the Pakistan health service perspective. Costings for the drugs, clinic, laboratory testing, staff and facility costs associated with each treatment regimen per patient will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent or sign consent forms with a fingerprint.
* Male or female, age ≥ 18 years.
* Willing to comply with study procedures
* Resident in the area and not planning to leave the region.
* Have a confirmed diagnosis at the time of screening of active hepatitis C infection - defined as detectable HCV RNA using a molecular diagnostic assay with a sensitivity of >100IU/ml OR detectable HCV Core antigen using an assay with a sensitivity of >1.5 pg/ml.
* Treatment experience within the last 24 months of antiviral therapy drugs recommended by the government program and administered in line with national recommendations. The current recommendations are that patients without cirrhosis should receive sofosbuvir 400 mg per day in combination with daclatasvir 60 mg per day for a total of 12 weeks and for patients with cirrhosis therapy should involve sofosbuvir 400 mg per day in combination with daclatasvir 60 mg per day for a total of 24 weeks. Patients who receive additional medication (including ribavirin) can be enrolled in the study but the additional medication should be noted.
* The subject's medical records must include sufficient detail of prior treatment to confirm eligibility.
* Have a stored sample of serum or plasma that is known to contain detectable HCV RNA and which can be made available to the study team or be willing to provide such a sample
* Have undergone, or be willing to undergo, an approved screening test for determining liver cirrhosis either by:

  1. APRI score - calculated from serum AST concentration in IU/L and platelet count /L (a result of ≥2 demonstrates presence of cirrhosis)
  2. Liver transient elastography assessment (a 'Fibroscan'). A result of ≥12.5 kPa will demonstrate cirrhosis.
  3. liver biopsy within 1 year of screening
* Females of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test on Day 1 prior to enrolment.
* Lactating females must agree to discontinue nursing before starting study drug.
* Subjects must be able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments.

Exclusion Criteria:

* Unwilling or unable to give consent
* Clinically significant illness (other than HCV) or other major medical condition that may interfere with the subject's treatment, assessment or compliance with protocol.
* History of discontinuation the most recent regime due to an adverse event
* Co-morbidities limiting life expectancy to less than 12 months
* Gastrointestinal disorder that could interfere with the absorption of the study drugs
* Significant cardiac disease
* Unstable psychiatric condition
* Significant drug allergy (e.g. hepatotoxicity)
* Infection with hepatitis B virus (HBV) or Human immunodeficiency virus (HIV)
* Unable or unwilling to undergo the necessary procedures - undergoing blood testing and ultrasound/fibroscan scanning.
* Previous poor compliance with medication (defined as failure to take >80% of the prescribed medication)
* Have undergone liver or other solid organ transplantation
* Have a current or recent diagnosis of hepatocellular carcinoma or any other malignancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Determine sustained virological response rate (SVR) | 36+/- 2 weeks from the point of randomisation
  Sustained virological response (SVR) defined as proportion of patients who are HCV RNA negative with a sensitive molecular test (sensitivity <100 IU/ml) 36 +/- 2 weeks from the time of randomisation.
  2. To determine the proportion of people with decompensated cirrhosis who achieve a sustained virological response (SVR) 36 weeks (+/-2 weeks) after first dose of medication (sofosbuvir/velpatasvir) administered.

SECONDARY OUTCOMES:
Cost effectiveness of treatment | 24 weeks after randomisation
  Cost-effectiveness analysis of retreatment with 12 or 24 week of sof/Vel compared to the standard of care of no re-treatment. Therefore, is it better to accept a lower success rate at lower cost or better to pay more for a few extra SVRs.
  We will measure the costs of treatment, lab tests, clinician/nurse team for the 12 and 24 week option and any standard of care disease monitoring (without treatment) and will include estimates of the costs of disease care for those not getting treated. We will measure health benefits in terms of DALYs averted or QALYs saved which will be estimated with a disease progression (and possibly transmission) model.
Health care costs | 24 weeks after randomisation
  To determine the health care costs associated with the different regimens in people with differing degrees of fibrosis.
Determine viral polymorphisms in HCV | 12 months
  To determine viral polymorphisms in HCV that are associated with a reduced response to antiviral therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Graham Foster, MBBS, Principal Investigator — Queen Mary University
Locations (1):
- Clinical trials unit, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] El-Akel W, El-Sayed MH, El Kassas M, El-Serafy M, Khairy M, Elsaeed K, Kabil K, Hassany M, Shawky A, Yosry A, Shaker MK, ElShazly Y, Waked I, Esmat G, Doss W. National treatment programme of hepatitis C in Egypt: Hepatitis C virus model of care. J Viral Hepat. 2017 Apr;24(4):262-267. doi: 10.1111/jvh.12668. Epub 2017 Feb 1. PMID 28145032
- [Result] Smith D, Magri A, Bonsall D, Ip CLC, Trebes A, Brown A, Piazza P, Bowden R, Nguyen D, Ansari MA, Simmonds P, Barnes E; STOP-HCV Consortium. Resistance analysis of genotype 3 hepatitis C virus indicates subtypes inherently resistant to nonstructural protein 5A inhibitors. Hepatology. 2019 May;69(5):1861-1872. doi: 10.1002/hep.29837. Epub 2018 Apr 27. PMID 29425396
- [Result] Lim AG, Walker JG, Mafirakureva N, Khalid GG, Qureshi H, Mahmood H, Trickey A, Fraser H, Aslam K, Falq G, Fortas C, Zahid H, Naveed A, Auat R, Saeed Q, Davies CF, Mukandavire C, Glass N, Maman D, Martin NK, Hickman M, May MT, Hamid S, Loarec A, Averhoff F, Vickerman P. Effects and cost of different strategies to eliminate hepatitis C virus transmission in Pakistan: a modelling analysis. Lancet Glob Health. 2020 Mar;8(3):e440-e450. doi: 10.1016/S2214-109X(20)30003-6. PMID 32087176
- [Result] Zeuzem S, Foster GR, Wang S, Asatryan A, Gane E, Feld JJ, Asselah T, Bourliere M, Ruane PJ, Wedemeyer H, Pol S, Flisiak R, Poordad F, Chuang WL, Stedman CA, Flamm S, Kwo P, Dore GJ, Sepulveda-Arzola G, Roberts SK, Soto-Malave R, Kaita K, Puoti M, Vierling J, Tam E, Vargas HE, Bruck R, Fuster F, Paik SW, Felizarta F, Kort J, Fu B, Liu R, Ng TI, Pilot-Matias T, Lin CW, Trinh R, Mensa FJ. Glecaprevir-Pibrentasvir for 8 or 12 Weeks in HCV Genotype 1 or 3 Infection. N Engl J Med. 2018 Jan 25;378(4):354-369. doi: 10.1056/NEJMoa1702417. PMID 29365309
- [Result] Foster GR, Afdhal N, Roberts SK, Brau N, Gane EJ, Pianko S, Lawitz E, Thompson A, Shiffman ML, Cooper C, Towner WJ, Conway B, Ruane P, Bourliere M, Asselah T, Berg T, Zeuzem S, Rosenberg W, Agarwal K, Stedman CA, Mo H, Dvory-Sobol H, Han L, Wang J, McNally J, Osinusi A, Brainard DM, McHutchison JG, Mazzotta F, Tran TT, Gordon SC, Patel K, Reau N, Mangia A, Sulkowski M; ASTRAL-2 Investigators; ASTRAL-3 Investigators. Sofosbuvir and Velpatasvir for HCV Genotype 2 and 3 Infection. N Engl J Med. 2015 Dec 31;373(27):2608-17. doi: 10.1056/NEJMoa1512612. Epub 2015 Nov 17. PMID 26575258
- [Result] Esteban R, Pineda JA, Calleja JL, Casado M, Rodriguez M, Turnes J, Morano Amado LE, Morillas RM, Forns X, Pascasio Acevedo JM, Andrade RJ, Rivero A, Carrion JA, Lens S, Riveiro-Barciela M, McNabb B, Zhang G, Camus G, Stamm LM, Brainard DM, Subramanian GM, Buti M. Efficacy of Sofosbuvir and Velpatasvir, With and Without Ribavirin, in Patients With Hepatitis C Virus Genotype 3 Infection and Cirrhosis. Gastroenterology. 2018 Oct;155(4):1120-1127.e4. doi: 10.1053/j.gastro.2018.06.042. Epub 2018 Jun 27. PMID 29958855
- [Result] Wing PAC, Jones M, Cheung M, DaSilva S, Bamford C, Jason Lee WY, Aranday-Cortes E, Da Silva Filipe A, McLauchlan J, Smith D, Irving W, Cunningham M, Ansari A, Barnes E, Foster GR. Amino Acid Substitutions in Genotype 3a Hepatitis C Virus Polymerase Protein Affect Responses to Sofosbuvir. Gastroenterology. 2019 Sep;157(3):692-704.e9. doi: 10.1053/j.gastro.2019.05.007. Epub 2019 May 10. PMID 31078622
- [Result] Huang R, Rao H, Xie Q, Gao Z, Li W, Jiang D, Mo H, Massetto B, Stamm LM, Brainard DM, Wei L. Comparison of the efficacy of sofosbuvir plus ribavirin in Chinese patients with genotype 3a or 3b HCV infection. J Med Virol. 2019 Jul;91(7):1313-1318. doi: 10.1002/jmv.25454. Epub 2019 Apr 3. PMID 30861150
- [Result] Lim AG, Qureshi H, Mahmood H, Hamid S, Davies CF, Trickey A, Glass N, Saeed Q, Fraser H, Walker JG, Mukandavire C, Hickman M, Martin NK, May MT, Averhoff F, Vickerman P. Curbing the hepatitis C virus epidemic in Pakistan: the impact of scaling up treatment and prevention for achieving elimination. Int J Epidemiol. 2018 Apr 1;47(2):550-560. doi: 10.1093/ije/dyx270. PMID 29309592

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-04-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT05248919/SAP_000.pdf